CLINICAL TRIAL: NCT04982341
Title: Effectiveness of High-flow Nasal Cannula and Prone Positioning in Awake Patients With COVID-19 and Severe Acute Respiratory Failure
Brief Title: HFNC and Prone Positioning in Awake Patients With Severe COVID-19
Status: Completed | Type: Observational
Sponsor: Hôpital Universitaire Fattouma Bourguiba (Other)
Responsible Party: Principal Investigator, Fekri Abroug, Professor Head of the ICU, Hôpital Universitaire Fattouma Bourguiba
Other Study IDs: FattoumaBourguiba_HFNC_Prone
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HFNC/prone: awake patients with COVID-19 and severe acute respiratory failure receiving HFNC in prone position
  Interventions: Procedure: prone position

INTERVENTIONS:
Procedure: prone position — patients are returned from prone to supine position while receiving oxygenation through HFNC

SUMMARY:
The investigators evaluate the effects of High-flow nasal cannula (HFNC) in association with prone in patients with Covid-19 severe ARF.

DETAILED DESCRIPTION:
The investigators evaluate the effects of High-flow nasal cannula (HFNC) in association with prone in patients with Covid-19 severe ARF.

All patients with ARF related to Covid-19 and admitted to the ICU are turned in prone position whenever tolerated, while receiving oxygenation with HFNC.

Outcomes of interest are the rate of success or failure (defined as the need for intubation and mechanical ventilation)

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years, admitted to the medical ICU for confirmed Covid-19 and acute hypoxemic respiratory failure

Exclusion Criteria:

* patients already intubated at admission or those requiring immediate intubation

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Covid-19 confirmed by rtPCR, suffering from acute hypoxemic failure requiring oxygenation
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Number of patients without intubation | through study completion, an average of 28 days
  successful oxygenation without intubation

CONTACTS AND LOCATIONS:
Overall Officials: Lamia Besbes, Prof, Study Chair — CPPRB
Locations (1):
- CHU F.Bourguiba, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No